CLINICAL TRIAL: NCT05100251
Title: An Open, Dose Escalation, Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of WBC100 in Patients with Advanced Solid Tumor
Brief Title: Clinical Trial of WBC100 on Advanced Solid Tumor
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Professor, Zhejiang University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WBC100
Record Dates: First submitted 2021-10-04; First posted 2021-10-29 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Solid Tumor
Keywords: C-myc; Solid tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Once every other day (QOD) (Experimental): (1) Once every other day (QOD): after a single-dose administration (C0) and 2-day washout period, subjects will start receiving multiple doses, for 2 consecutive weeks, followed by a 1-week rest period, with 3 weeks as one treatment cycle
  Interventions: Drug: WBC100 QOD
- Twice daily (BID) (Experimental): (2) Twice daily (BID): dosing for 2 consecutive weeks, followed by a 1-week rest period, with 3 weeks as one treatment cycle;
  Interventions: Drug: WBC100 BID
- Once daily (QD) (Experimental): Once daily (QD): dosing 3 consecutive weeks (with QD dosing for the first 5 days of each week followed by a 2-day rest), followed by a 1-week rest period, with a 4 weeks as one cycle
  Interventions: Drug: WBC100 QD

INTERVENTIONS:
Drug: WBC100 QOD — The first stage: single dose escalation according to classic "3+3" dose escalation method. 7 increasing dose levels were set up, with 3 to 6 cases per dose. The first dose group is 0.5 mg QOD. The second dose group is 1mg QOD. The third dose group is 1.5 mg QOD. The fourth dose group is 2.0 mg QOD. The fifth dose group is 2.5 mg QOD. The sixth dose group is 3.0 mg QOD. The seven dose group is 3.5 mg QOD. In each dose group, patients take WBC100 once on cycle 0. After a washout period of 2 days, patents start subsequent 4 weeks cycles until progression disease or intolerable toxicity. In each cycle, patient was on WBC100 every for 3 weeks and off for 1 week.
  The second stage: Two dose levels will be chosen according to data from the first stage. Each dose stage will enroll 12 c-myc-positive patients with a selected cancer type
  Arms: Once every other day (QOD)
Drug: WBC100 QD — The first stage: single dose escalation according to classic "3+3" dose escalation method. 6 increasing dose levels were set up, with 3 to 6 cases per dose. The first dose group is 0.5 mg QD. The second dose group is 1mg QD. The third dose group is 1.5 mg QD. The fourth dose group is 2.0 mg QD. The fifth dose group is 2.5 mg QD. The sixth dose group is 3.0 mg QD. In each dose group, the patient was on WBC100 until progression disease or intolerable toxicity. Patient was on WBC100 every for for 3 consecutive weeks (with QD dosing for the first 5 days of each week followed by a 2-day rest), followed by a 1-week rest period, with a 4 weeks as one cycle. The second stage: Two dose levels will be chosen according to data from the first stage. Each dose stage will enroll 12 c-myc-positive patients with a selected cancer type
  Arms: Once daily (QD)
Drug: WBC100 BID — The first stage: single dose escalation according to classic "3+3" dose escalation method. 4 increasing dose levels were set up, with 3 to 6 cases per dose. The first dose group is 0.5 mg QD. The second dose group is 1mg QD. The third dose group is 1.5 mg QD. The fourth dose group is 2.0 mg QD. In each dose group, the patient was on WBC100 until progression disease or intolerable toxicity. Patient was on WBC100 every for 2 consecutive weeks, followed by a 1-week rest period, with 3 weeks as one treatment cycle; The second stage: Two dose levels will be chosen according to data from the first stage. Each dose stage will enroll 12 c-myc-positive patients with a selected cancer type
  Arms: Twice daily (BID)

SUMMARY:
This is a phase I clinical study of WBC100 in Patients with advanced solid tumor.

DETAILED DESCRIPTION:
This is a phase I open-label, single and dose escalation study to evaluate the safety, pharmacokinetics, and preliminary efficacy of WBC100, a drug targeting c-myc, in subjects who have been diagnosed with c-myc positive advanced solid tumor and refractory or intolerant to current standard systemic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent, able to follow protocol requirements；
2. Aged 18 to 75 years, male or female
3. （1）Dose escalation stage: Histopathology or cytology proven patients with advanced solid tumor with positive C-myc expression who have developed progressive disease or intolerability after at least one line of standard systemic therapies.（2）Dose expansion stage: Histopathology or cytology proven patients with advanced solid tumor of a selected cancer type with positive C-myc expression who have developed progressive disease or intolerability after at least one line of standard systemic therapies. Positive C-myc refers to more than 1% tumor cells are detected 1+ by immunohistochemistry (IHC) in histologic section.
4. ECOG Performance Status score: 0 to 2 points
5. Expected survival is > 3 months
6. Adequate hematologic and organ functions (without persistent supportive treatment)

   1. Absolute Neutrophil Count > 1.5 × 109/L, Platelet count ≥ 75 × 109/L, Hemoglobin > 8.5 g/dL
   2. INR and PT ≤ 2 × ULN
   3. ALB > 3.0 g/dL, Bilirubin level ≤ 2 × ULN, AST and ALT ≤ 2 × ULN or < 5 × ULN in the presence of liver metastases
   4. Calculated creatinine clearance (e.g. Cockcroft-Gault) ≥ 60 ml/min or serum creatinine ≤ 1.5 × ULN

   f. Left ventricular ejection fraction (LVEF) ≥ 50%. Heart rate (HR) ≥ 60 bpm. QT intervals, male ≤ 450 ms, female ≤ 470 ms
7. According to RECIST 1.1, patients have at least one evaluable target lesion(only for dose expansion stage)
8. Female patients of child-bearing potential or male subjects whose spouses are women of childbearing potential must agree to use a reliable method of contraception (IUD, oral contraceptive, condom) throughout the treatment period and for 3 months after discontinuation of WBC100. Female patients of child-bearing age must undergo a serum pregnancy test before the initiation of the study and the result must be negative.

Exclusion Criteria:

1. Allergic to WBC100 or its excipients or with allergic constitution
2. Major surgery, active ulcer or unhealing wound occurred within 4 weeks before first dose
3. Taken drugs in other clinical trials within 4 weeks or still in the safety follow-up period
4. Subjects have Spinal compression, brain metastases and meningeal metastases (subjects who is asymptomatic, stable or with no need for steroid for at least 4 weeks before first dose are allowed)
5. Subjects have history of cardiac insufficiency (NYHA III-IV) or uncontrolled congestive heart failure (NYHA II-IV) within 6 months before consent
6. Subjects have risk factors of QT intervals prolongation or arrhythmia, such as Idiopathic Q-T interval prolongation syndrome or history of drug induced arrhythmia
7. Subject have any condition within 6 months before consent: unstable angina pectoris requiring surgical intervention, uncontrolled hypertension (systolic pressure ≥ 140 mmHg, diastolic pressure ≥ 90 mmHg), myocardial infarction, stroke (lacunar infarction is allowed), Coronary/peripheral artery bypass surgery, pulmonary embolism
8. Infection of HIV, active infection of HBV (HBV DNA > 1000 IU/ml) active infection of HC (HCV-RNA ≥ upper limits of normal)
9. History of severe infection within 28 days before enrolled, including uncontrolled infection requiring systemic treatment of bacteria, virus and fungus
10. The side effects caused by the previous treatment of the subjects did not return to grade ≤1 according to CTCAE 5.0 with exception of tolerable events determined by investigator such as hair loss and grade 2 Peripheral neuropathy
11. Subjects with uncontrolled nausea or vomiting, chronic gastrointestinal diseases, unable to swallow pills, enterostomy, uncontrolled diarrhea or any intestinal surgery that cause insufficient absorption of WBC100
12. Subjects taking any strong CYP inducers or inhibitors or Chinese medicine within 7 days prior to the first dose of study drug
13. History of malignancy in the last 2 years with the exception of patients with prior history of in situ breast cancer, in situ cervical cancer, basal or squamous cell skin cancer who have already been cured
14. Subjects who have antitumor therapy within 28 days prior to first dose of WBC100, such as monoclonal antibody, chemotherapy, radiotherapy and Chinese medicine
15. Subjects have mental disorders or history of drug abuse that may limit subjects' participation in this trial
16. Unable to tolerate intravenous blood collection
17. According to the investigators' evaluation, patients are unable or unwilling to comply with the requirements of the study protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2025-10-25 (Estimated); Study Completion 2025-10-25 (Estimated)

PRIMARY OUTCOMES:
Frequency of Adverse Event and Severe Adverse Event | 2 years
  AEs and SAEs will be assessed by CTCAE v5.0
Dose limited toxicity（DLT） | 28 days
  safety
Maximum Tolerated Dose（MTD） | 28 days
  The highest dose level at which < 2 of 6 subjects experienced a dose limiting toxicity during the first 28 days of the treatment period

SECONDARY OUTCOMES:
Cmax | 28 days
  Peak plasma concentration after one dose
Tmax | 28 days
  Time to peak plasma concentration after one dose
AUC0-t | 28 days
  Area under the plasma concentration versus time curve after one dose and multiple dose；time range from 0 to last point when plasma concentration is detectable
AUC0-inf | 28 days
  Area under the plasma concentration versus time curve；time range from 0 to infinity
T1/2 | 28 days
  half-life period
λz | 28 days
  elimination rate constant
CL/F | 28 days
  apparent clearance
Vz/F | 28 days
  apparent volume of distribution
Cmax, ss | 28 days
  Steady peak plasma concentration after multiple dose
Cmin, ss | 28 days
  Steady minimal plasma concentration after multiple dose
Cavg | 28 days
  Steady averagel plasma concentration after multiple dose
Tmax, ss | 28 days
  Time to steady peak plasma concentration after multiple dose
CLss/F | 28 days
  steady apparent clearance
Vss/F | 28 days
  steady apparent volume of distribution
ARCmax | 28 days
  Peak concerntration cumulative coefficient
ARAUC | 28 days
  AUC cumulative coefficient
DF | 28 days
  degree of fluctuation
CA19-9 | 28 days
  Change of CA19-9
CA125 | 28 days
  Change of CA125
Serum ferritin | 28 days
  change of serum ferritin
Progression-free survival (PFS) | 2 years
  The period from the day when the subject receives the first study treatment to the first recorded tumor progression (whether treated or not) or death of any cause, which occurs first
Duration of response (DOR) | 2 years
  The period from the first evaluation of complete response ( CR) or partial response (PR) to the first evaluation of progressive disease (PD)or death of any cause
Objective response rate (ORR) | 2 years
  The number of cases in which tumor size is reduced to partial response (PR) or complete response (CR) / the total number of evaluable cases (%). In the event of partial response( PR) or complete response (CR), the subjects should confirm it no less than 4 weeks after the first evaluation
change of tumor size | 52 weeks
  The major axis change of target lesion relative to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Tingbo Liang, Principal Investigator — Zhejiang University
Locations (1):
- the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No